CLINICAL TRIAL: NCT04979962
Title: Colorectal Polyp Detection Comparing Computer Assisted Colonoscopy With Conventional Colonoscopy
Brief Title: AI Colorectal Polyp Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujifilm Medical Systems USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: P-21-006
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Polyp Colorectal; Adenoma Colon

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be randomized 1:1, inspection with computer assisted colonoscopy: inspection with conventional colonoscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- CAC Group (Experimental): Inspection with computer assisted colonoscopy.
  Interventions: Device: EW10-EC02 (Endoscopy Support Program)
- CC Group (No Intervention): Inspection with conventional colonoscopy

INTERVENTIONS:
Device: EW10-EC02 (Endoscopy Support Program) — EW10-EC02 is intended to automatically detect the location of suspected polyps in colonoscopy exams. Identified polyps are highlighted to the clinician in real-time during the exam, as a video image superimposed on the endoscope monitor. EW10-EC02 is limited to the detection of suspected findings, and should not be used in lieu of full patient evaluation or relied upon to make or confirm a diagnosis.
  Arms: CAC Group

SUMMARY:
This study is intended to demonstrate the superiority of colorectal polyp detection using computer-assisted colonoscopy compared to conventional colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Average risk subjects undergoing their first colonoscopy (screening) or follow-up colonoscopy for previous history of polyps (surveillance interval of 3 years or greater)
* Patients aged 45 or older
* Patients who can provide an informed consent

Exclusion Criteria:

* Patients with history of colon resection, Inflammatory Bowel Disease (IBD), Familial Adenomatous Polyposis (FAP), severe comorbidity, including end-stage cardiovascular/pulmonary/liver/renal disease
* Patients who are pregnant or are planning pregnancy during study period
* Patients who are not able to or refuse to give informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1162 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Adenoma per colonoscopy (APC) | 1 day/procedure
  Total number of histologically confirmed adenomas and carcinomas detected in the colonoscopy divided by the total number of colonoscopies

SECONDARY OUTCOMES:
Positive predictive value (PPV) | 1 day/procedure
  Total number of histologically confirmed adenomas and carcinomas detected during the colonoscopy, divided by the total number of excisions in the colonoscopy
Adenoma detection rate (ADR) | 1 day/procedure
  proportion of patients with at least one histologically confirmed adenoma or carcinoma detected in the colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, MD, Principal Investigator — Kansas City VA Medical Center
Locations (10):
- United States (10):
  - Keck Medicine University of Southern California, Los Angeles, California
  - Largo Medical Center (HCA), Largo, Florida
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - GI Associates, Flowood, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Kansas City VA Medical Center, Kansas City, Missouri
  - New York University/Manhattan Endoscopy, New York, New York
  - Columbia University Medical Center, New York, New York
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Desai M, Ausk K, Brannan D, Chhabra R, Chan W, Chiorean M, Gross SA, Girotra M, Haber G, Hogan RB, Jacob B, Jonnalagadda S, Iles-Shih L, Kumar N, Law J, Lee L, Lin O, Mizrahi M, Pacheco P, Parasa S, Phan J, Reeves V, Sethi A, Snell D, Underwood J, Venu N, Visrodia K, Wong A, Winn J, Wright CH, Sharma P. Use of a Novel Artificial Intelligence System Leads to the Detection of Significantly Higher Number of Adenomas During Screening and Surveillance Colonoscopy: Results From a Large, Prospective, US Multicenter, Randomized Clinical Trial. Am J Gastroenterol. 2024 Jul 1;119(7):1383-1391. doi: 10.14309/ajg.0000000000002664. Epub 2024 Jan 18. PMID 38235741